CLINICAL TRIAL: NCT03311217
Title: Tribal Health and Resilience in Vulnerable Environments
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HL117729 (NIH)
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial with four communities assigned to intervention and four communities assigned to control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Healthy retail strategies will be implemented in tribally owned convenience stores in these communities. Specific strategies include pricing discounts, promotional signage, incorporation of new product, and placement of healthier items on shelves.
  Interventions: Behavioral: Healthy retail strategies
- Control group (No Intervention): No intervention will be implemented in the stores in the control communities.

INTERVENTIONS:
Behavioral: Healthy retail strategies
  Arms: Intervention group

SUMMARY:
The THRIVE study is a healthy retail intervention that improves the food environments in tribally owned and operated convenience stores in the Chickasaw Nation and Choctaw Nation of Oklahoma.

DETAILED DESCRIPTION:
The THRIVE study is a cluster randomized trial, using a community-based participatory research approach, of "healthy makeovers" in eight convenience stores owned and operated by the Chickasaw Nation and Choctaw Nation of Oklahoma. The study will test the ability of tribal nations to increase fruit and vegetable purchasing and consumption among tribal members through environmental and policy approaches. Investigators hypothesize that tribal members exposed to the highest doses of the intervention (i.e. those who visit the intervention convenience stores the most) will increase their fruit and vegetable intake. Individual-level changes in fruit and vegetable intake will be measured via a survey administered to a cohort of 1600 American Indian shoppers before and after the intervention. A multimedia manual, Website, and documentary film will be created as part of the implementation of THRIVE to engage tribal citizens, enhance local knowledge, and guide other tribes to improve their food and physical activity environments.

ELIGIBILITY:
Inclusion criteria

* American Indian or Alaska Native
* Residing in the tribal jurisdictional areas
* No plans of moving within 12 months
* Self-report shopping at the stores for food at least 3 times per week

Exclusion Criteria:

• Anyone who does not meet these criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1634 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Fruit intake | 9 to 12months duration depending on tribe and store
  Self reported via 6 questions asking about consumption of intervention foods
Vegetable intake | 9 to 12months duration depending on tribe and store
  Self reported via 6 questions asking about consumption of intervention foods

CONTACTS AND LOCATIONS:
Overall Officials: Valarie Jernigan, DrPH, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jernigan VBB, Wetherill M, Hearod J, Jacob T, Salvatore AL, Cannady T, Grammar M, Standridge J, Fox J, Spiegel J, Wiley A, Noonan C, Buchwald D. Cardiovascular Disease Risk Factors and Health Outcomes Among American Indians in Oklahoma: the THRIVE Study. J Racial Ethn Health Disparities. 2017 Dec;4(6):1061-1068. doi: 10.1007/s40615-016-0310-4. Epub 2016 Dec 6. PMID 27924618
- [Background] Blue Bird Jernigan V, Wetherill MS, Hearod J, Jacob T, Salvatore AL, Cannady T, Grammar M, Standridge J, Fox J, Spiegel J, Wiley A, Noonan C, Buchwald D. Food Insecurity and Chronic Diseases Among American Indians in Rural Oklahoma: The THRIVE Study. Am J Public Health. 2017 Mar;107(3):441-446. doi: 10.2105/AJPH.2016.303605. Epub 2017 Jan 19. PMID 28103070